CLINICAL TRIAL: NCT03429426
Title: An Observational Study of Bone Erosion Determination and Progression in Rheumatoid Arthritis Assessed by HR-pQCT and Conventional X-ray
Brief Title: Progression of Bone Erosions in Rheumatoid Arthritis Assessed by HR-pQCT and Conventional X-ray
Acronym: RACTX
Status: Enrolling by invitation | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Rasmus Klose-Jensen, MD, PhD Student, Aarhus University Hospital
Other Study IDs: RACTX
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; High-resolution peripheral quantitative computed tomography; Radiography
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A research biobank for blood samples will be established for the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis: Patients with Rheumatoid arthritis ≥5 years according to the ACR/EULAR 2010 classification criteria or the American Rheumatism Association 1987 revised criteria.
  ICD-10: M059 Seropositive rheumatoid arthritis UNS, M060 Seronegative rheumatoid arthritis, M069 Rheumatoid arthritis UNS.
- Pre-Rheumatoid arthritis: Patients with joint pain, but no swelling and Anti-CCP 3 times above the upper limit.
- Healthy Subjects: Healthy age- and sex-matched Individuals are recruited, as a control group.

SUMMARY:
Today, regular X-ray examination is not sufficiently sensitive for detecting progression of bone destruction in rheumatoid arthritis, but a new type of high-resolution CT scanner, the High-Resolution peripheral Quantitative Computed Tomography (HR-pQCT) can detect very early and minor joint injuries.

The purpose of this study is to use HR-pQCT techniques to look at the damage and disease activity progression in the hand and wrist joints of patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The design of the trial is an observational study with three distinct groups. At the start of the trial period and at one-year of follow-up, the trial subject will have their hand X-rayed by conventional radiography, and their metacarpophalangeal (MCP) joint and wrist scanned by HR-pQCT-Imaging. The 28-joint Disease Activity Score(DAS28-CRP), Health Assessment Questionnaire (HAQ), Visual analogue scale(VAS)-score for pain, fatigue and quality of life are performed to investigate the correlation between radiographic changes and disease activity. Blood samples are collected to investigate serological markers of bone metabolism and inflammation and the radiographic changes. The following groups are investigated:

* Rheumatoid Arthritis(RA): Patients with RA ≥5 years according to the ACR/EULAR 2010 classification criteria or the American Rheumatism Association 1987 revised criteria are recruited from the outpatient clinic at the Department of Rheumatology, Aarhus University Hospital. Treatment will be adjusted according to the patient's need and according to national guidelines. (n=450)
* Pre-RA patients: Patients with pre-RA, (joint pain, but no swelling and Anti-CCP 3 times above the upper limit) are recruited from the outpatient clinic at the Department of Rheumatology, Aarhus University Hospital. (n=75)
* Healthy subjects: Healthy age- and sex-matched Individuals are recruited, as a control group, by posting at libraries in Aarhus, Aarhus University, Aarhus University Hospital and postings on the websites www.forsøgsperson.dk and www.Sundhed.dk. (N=100)

ELIGIBILITY:
Rheumatoid arthritis patients Inclusion criteria

* Patients (> 18 years) with rheumatoid arthritis ≥5 years according to the ACR/EULAR (2010) classification criteria or American Rheumatism Association 1987 revised criteria for the patients who were diagnosed before 2010.
* Patients who are receiving treatment on an outpatient basis.
* Ability and willingness to give written informed consent and to meet the requirements of the trial protocol.

Exclusion criteria

* Patients who have previously suffered trauma in the form of fracture or luxation of the hand are excluded.
* Evidence of active malignant disease.
* Hypo- or hyperthyroidism.
* Hypocalcaemia.
* Impaired renal function (eGFR <35ml/min).
* Pregnancy. Pre-rheumatoid arthritis patients Inclusion criteria
* Age over 18 years.
* Anti-CCP 3 times the upper limit of the reference interval.
* Arthralgia.
* Ability and willingness to give written informed consent and to meet the requirements of the trial protocol.

Exclusion criteria

* Pregnancy.
* Swelling of joints. Verified by clinical ultrasound.
* Patients who have previously suffered trauma in the form of fracture or luxation of the hand are excluded.
* Evidence of malignant disease.
* Hypo- or hyperthyroidism.
* Hypocalcaemia. Healthy subjects Inclusion criteria
* Age over 18 years.
* No joint complaints.
* Ability and willingness to give written informed consent and to meet the requirements of the trial protocol.

Exclusion criteria

* Patients who have previously suffered trauma in the form of fracture or luxation of the hand are excluded.
* Evidence of malignant disease.
* Hypo- or hyperthyroidism.
* Hypocalcaemia.
* Impaired renal function (eGFR <35ml/min).
* Earlier or present rheumatological disease or bone metabolic disease.
* Positive anti-CCP.
* Pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients and pre-rheumatoid patients are recruited from the outpatient clinic at the Department of Rheumatology, Aarhus University Hospital.
  Healthy age- and sex-matched Individuals are recruited, as a control group, by posting at libraries in Aarhus, Aarhus University, Aarhus University Hospital and postings on the websites www.forsøgsperson.dk and www.Sundhed.dk.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Erosion changes by HR-pQCT | One year
  Changes in bone erosions volume in mm3 by HR-pQCT-imaging from baseline to one-year follow-up, in the three groups.
Volumetric bone mineral density(vBMD) changes by HR-pQCT | One year
  Changes in volumetric bone mineral density(vBMD) in mgHA/cm3 by HR-pQCT-imaging from baseline to one-year follow-up, in the three groups.
Erosion changes by HR-pQCT | One year
  Changes in bone erosions width in mm by HR-pQCT-imaging from baseline to one-year follow-up, in the three groups.
Erosion changes by HR-pQCT | One year
  Changes in bone erosions depth in mm by HR-pQCT-imaging from baseline to one-year follow-up, in the three groups.

SECONDARY OUTCOMES:
Radiographic erosion score | One year
  Change in Sharp/van der Heijde (SvH) score from baseline to one-year follow-up, in the three groups.
CTX | one year
  Changes from baseline to one-year follow-up in C-terminal telopeptide (CTX) in pg/mL, in the three groups.
P1NP | one year
  Changes from baseline to one-year follow-up in Procollagen type 1 N-terminal propeptide (P1NP) in pg/mL, in the three groups.
BAP | one year
  Changes from baseline to one-year follow-up in Bone-specific alkaline phosphatase (BAP) in pg/mL, in the three groups.
TNF-α | one year
  Changes from baseline to one-year follow-up in the Tumor necrosis factor-alfa (TNF-α) in pg/mL, in the three groups.
RANK-L | one year
  Changes from baseline to one-year follow-up in RANK-Ligand (RANK-L) in pg/mL, in the three groups.
OPG | one year
  Changes from baseline to one-year follow-up in Osteoprotegerin (OPG) in pg/mL, in the three groups.
BGLAP | one year
  Changes from baseline to one-year follow-up in Osteocalcin (BGLAP) in pg/mL, in the three groups.
SCL | one year
  Changes from baseline to one-year follow-up in Sclerostin(SCL) in pg/mL, in the three groups.
Dkk-1 | one year
  Changes from baseline to one-year follow-up in Dickkopf-related protein 1 (Dkk-1) in pg/mL, in the three groups.
IL-1 | one year
  Changes from baseline to one-year follow-up in Interleukins 1 (IL-1) in pg/mL, in the three groups.
IL-6 | one year
  Changes from baseline to one-year follow-up in Interleukins 6 (IL-6) in pg/mL, in the three groups.
IL-15 | one year
  Changes from baseline to one-year follow-up in Interleukins 15 (IL-15) in pg/mL, in the three groups.
IL-16 | one year
  Changes from baseline to one-year follow-up in Interleukins 16 (IL-16) in pg/mL, in the three groups.
IL-17 | one year
  Changes from baseline to one-year follow-up in Interleukins 17 (IL-17) in pg/mL, in the three groups.
IL-22 | one year
  Changes from baseline to one-year follow-up in Interleukins 22 (IL-22) in pg/mL, in the three groups.
IL-33 | one year
  Changes from baseline to one-year follow-up in Interleukins 33 (IL-33) in pg/mL, in the three groups.
CCL11 | one year
  Changes from baseline to one-year follow-up in Chemokine ligand 11 (CCL11) in pg/mL, in the three groups.
CXCL13 | one year
  Changes from baseline to one-year follow-up in Chemokine (C-X-C) motif ligand (CXCL13) in pg/mL, in the three groups.
TRACP 5b | one year
  Changes from baseline to one-year follow-up in Tartrate-resistant acid phosphatase 5b (TRACP 5b) in pg/mL, in the three groups.
CRP | one year
  Changes from baseline to one-year follow-up in C-reactive protein (CRP) in mg/L, in the three groups.
Disease Activity Score | one year
  Disease Activity Score (DAS28-CRP) [2.0-10.0]
Health Assessment Questionnaire | one year
  Health Assessment Questionnaire (HAQ) [0-3 HAQ Total Score]
VAS for pain | one year
  Visual Analog Scale(VAS) for pain [0-100mm]
VAS for fatigue | one year
  Visual Analog Scale(VAS) for fatigue [0-100mm]
VAS for quality of life | one year
  Visual Analog Scale(VAS) for quality of life [0-100mm]

OTHER OUTCOMES:
areal bone mineral density (aBMD) | one year
  aBMD in the lumbar spine, and the left hip by DXA, in RA patients

CONTACTS AND LOCATIONS:
Overall Officials: Ellen-Margrethe Hauge, MD, PhD, Study Director — Department of Rheumatology - Aarhus University Hospital
Locations (1):
- Department of Rheumatology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Therkildsen J, Klose-Jensen R, Langdahl B, Bruel A, Thomsen JS, Moger C, Stilling M, Keller KK, Hauge EM. Mapping the bare area and transcortical pores in finger joints: co-location with bone erosions in rheumatoid arthritis. RMD Open. 2026 Jan 22;12(1):e006371. doi: 10.1136/rmdopen-2025-006371. PMID 41571324
- [Derived] Therkildsen J, Klose-Jensen R, Hanel M, Langdahl BL, Thomsen JS, Manske SL, Keller KK, Hauge EM. Detecting new erosions in rheumatoid arthritis over one year - Radiography and high-resolution computed tomography of finger joints. Joint Bone Spine. 2025 Jan;92(1):105812. doi: 10.1016/j.jbspin.2024.105812. Epub 2024 Nov 14. PMID 39547428
- [Derived] Klose-Jensen R, Therkildsen J, Blavnsfeldt AG, Langdahl BL, Zejden A, Thygesen J, Keller KK, Hauge EM. Diagnostic accuracy of high-resolution peripheral quantitative computed tomography and X-ray for classifying erosive rheumatoid arthritis. Rheumatology (Oxford). 2022 Mar 2;61(3):963-973. doi: 10.1093/rheumatology/keab446. PMID 34015091

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03429426/Prot_SAP_000.pdf